CLINICAL TRIAL: NCT04429906
Title: Evaluation of Accuracy of Blood Oxygen Saturation Detection Function of Huami Smart Wearable Device
Brief Title: Diagnostic Study of Huami Smart Wearable Device
Acronym: DSHWD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Anhui Huami Information Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Guangfa Wang, Professor & MD., Peking University First Hospital
Other Study IDs: 2020114-0604
Record Dates: First submitted 2020-06-04; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Oxygen Saturation
Keywords: Oxygen saturation Smart wearable device Accuracy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- test group: Wear the pulse-oxygen monitoring finger set of the medical monitor while wearing the Huami Smart Wearable device on the ipsilateral wrist according to the instructions for use. The medical monitor displays a steady pulse oximetry level for at least 30 seconds, starts the first measurement, slides the main dial page of the wearable device to the "Oxygen Saturation" measurement interface, clicks the measurement button to start the single measurement of blood oxygen saturation. Record the pulse oximetry and pulse rate values measured at the same time by the medical monitor and the Huami Smart Wearable Pulse Oximetry Device, respectively. After an interval of 30 seconds, repeat the above steps to start the second measurement and record the measured value. After an interval of 30 seconds, repeat the above steps to start the third measurement and record the measured value. The average of three measurements was taken as data for the test group.
  Interventions: Device: Huami smart wearable device
- control group A: Pulse oximetry monitor/desktop ECG monitor with a medical device registration certificate was selected as reference device A. The mean value of qualified pulse oximetry measured by pulse oximetry monitor/desktop ECG monitor within 2 minutes of each successive measurement of the Huami Smart Wearable Device was used as control group A measurement.
- control group B: A carbon monoxide blood gas analyzer (CO-oximeter) was selected as reference device B. Arterial blood was sampled and arterial oxygen saturation (SaO2) was obtained from the blood gas analyzer as a control group B measurement.

INTERVENTIONS:
Device: Huami smart wearable device — Wear the pulse-oxygen monitoring finger set of the medical monitor while wearing the Huami Smart Wearable device on the ipsilateral wrist according to the instructions for use. The medical monitor displays a steady pulse oximetry level for at least 30 seconds, starts the first measurement, slides the main dial page of the wearable device to the "Oxygen Saturation" measurement interface, clicks the measurement button to start the single measurement of blood oxygen saturation. Record the pulse oximetry and pulse rate values measured at the same time by the medical monitor and the Huami Smart Wearable Pulse Oximetry Device, respectively. After an interval of 30 seconds, repeat the above steps to start the second measurement and record the measured value. After an interval of 30 seconds, repeat the above steps to start the third measurement and record the measured value. The average of three measurements was taken as data for the test group.
  Groups: test group

SUMMARY:
This is a cross-sectional diagnostic study. In this study, wrist oxygen saturation (SwO2) will be measured by Huami smart wearable device, SpO2 of pulse oxygen saturation monitor with medical device registration certificate and SaO2 of arterial blood gas analysis will be used as reference values. A total of 180 group data will be measured in 30~50 patients with SaO2/ SpO2 between 80%∽100%. The investigators aim to evaluate the accuracy of blood oxygen saturation detection function of huami smart wearable device.

DETAILED DESCRIPTION:
This is a cross-sectional diagnostic study. 30~50 inpatient aged 18～85y with SaO2/ SpO2 between 80%∽100% will be recruited from the Department of Respiratory and Critical Care of Peking University First Hospital. 180 group data ( 37 of SaO2/ SpO2 between 80%∽90%, 143 of SaO2/ SpO2 between 90%∽100%) will be measured, with an average of 4-6 groups per patient. Some clinical information such as demographic data, laboratory tests, comorbidity, smoking habit and will be collected. Patients have their pulse oximetry measured multiple times using a pulse oximeter/tabletop electrocardiograph with a medical device registration certificate, and arterial blood gas analysis will be performed if required. While monitoring the pulse oximetry, a Huami smart wearable device is worn on the ipsilateral wrist to determine blood oxygen saturation. Primary outcome is the wearable device oximetry accuracy Arms (root mean square value of the SwO2-RefSpO2 difference) using a medical device registration certificate pulse oximetry monitor/tabletop ECG monitor as a reference..

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2020-114). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients in the Department of Respiratory and Critical Care at Peking University First Hospital
2. Oxygen intake or no oxygen intake when enrolled: 80%≤SaO2/SpO2≤100%
3. Age between 18 and 85 years, either gender
4. COHb<3%, MetHb<2%;
5. Sign an informed consent or sign an informed consent by a legally authorized representative;
6. Be willing and able to follow the research program.

Exclusion Criteria:

1. current smokers or those exposed to high levels of carbon monoxide.
2. critically ill patients who are in a state of shock, resulting in peripheral circulation disorders.
3. Patients with hypothermia below 35°C.
4. Patients with bilateral wrist and hand oedema, soft tissue damage to the wrist, skin incomplete and unable to wear a watch/ bracelet.
5. Vascular blood supply abnormalities of both upper limbs (occlusion, thrombosis, post-trauma, etc.), which affects the test results
6. Patients with bilateral upper extremity pigmentation affecting the test results;
7. Patients with limb mobility impairment due to severe cerebrovascular disease sequelae.
8. Patients with severe mental system disease that makes it impossible to cooperate with the researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients in the Department of Respiratory and Critical Care at Peking University First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Wearable device oximetry accuracy Arms | 30mins
  Record the pulse oximetry and pulse rate values measured at the same time by the medical monitor and the Huami Smart Wearable Pulse Oximetry Device, respectively. After an interval of 30 seconds, repeat the above steps to start the second measurement and record the measured value. After an interval of 30 seconds, repeat the above steps to start the third measurement and record the measured value. The average of three measurements was taken as data for the test group.
  Pulse oximetry monitor/desktop ECG monitor with a medical device registration certificate was selected as reference device A. The mean value of qualified pulse oximetry measured by pulse oximetry monitor/desktop ECG monitor was used as control group A measurement.
  Wearable device oximetry accuracy Arms (root mean square value of the SwO2-RefSpO2 difference) using a medical device registration certificate pulse oximetry monitor/tabletop ECG monitor as a reference.

SECONDARY OUTCOMES:
Wearable device blood oxygen saturation accuracy Arms | 30mins
  Record the pulse oximetry and pulse rate values measured by the Huami Smart Wearable Pulse Oximetry Device. After an interval of 30 seconds, repeat the above steps to start the second measurement and record the measured value. After an interval of 30 seconds, repeat the above steps to start the third measurement and record the measured value. The average of three measurements was taken as data for the test group.A carbon monoxide blood gas analyzer (CO-oximeter) was selected as reference device B. Arterial blood was sampled and arterial oxygen saturation (SaO2) was obtained from the blood gas analyzer as a control group B measurement.Wearable device blood oxygen saturation accuracy Arms (expressed as root mean square value of the SwO2-SaO2 difference) using a carbon monoxide - blood gas analyzer (CO-oximeter) as reference.
Accuracy of blood oxygen saturation of wearable devices when SpO2/SaO2 is at 90%-100%. | 30mins
  When SpO2/SaO2 is at 90%-100%,wearable device oximetry accuracy Arms (root mean square value of the SwO2-RefSpO2 difference) using a medical device registration certificate pulse oximetry monitor/tabletop ECG monitor as a reference;wearable device blood oxygen saturation accuracy Arms (expressed as root mean square value of the SwO2-SaO2 difference) using a carbon monoxide - blood gas analyzer (CO-oximeter) as reference.
Accuracy of blood oxygen saturation of wearable devices when SpO2/SaO2 is at 80%-89%. | 30mins
  when SpO2/SaO2 is at 80%-89%,wearable device oximetry accuracy Arms (root mean square value of the SwO2-RefSpO2 difference) using a medical device registration certificate pulse oximetry monitor/tabletop ECG monitor as a reference;wearable device blood oxygen saturation accuracy Arms (expressed as root mean square value of the SwO2-SaO2 difference) using a carbon monoxide - blood gas analyzer (CO-oximeter) as reference.
Correlation analysis of parameters that have an impact on the accuracy of blood oxygen saturation of wearable devices. | 30mins
  When the test result is negative, evaluate the parameters that have an impact on the accuracy of blood oxygen saturation of wearable devices.
The variability of blood oxygen saturation of wearable devices tested three times. | 30mins
  Record the pulse oximetry and pulse rate values measured at the same time by the medical monitor and the Huami Smart Wearable Pulse Oximetry Device, respectively. After an interval of 30 seconds, repeat the above steps to start the second measurement and record the measured value. After an interval of 30 seconds, repeat the above steps to start the third measurement and record the measured value. Evaluate the variability of blood oxygen saturation of wearable devices tested three times.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olsen M, Zeitzer JM, Richardson RN, Davidenko P, Jennum PJ, Sorensen HBD, Mignot E. A Flexible Deep Learning Architecture for Temporal Sleep Stage Classification Using Accelerometry and Photoplethysmography. IEEE Trans Biomed Eng. 2023 Jan;70(1):228-237. doi: 10.1109/TBME.2022.3187945. Epub 2022 Dec 26. PMID 35786544